CLINICAL TRIAL: NCT03809143
Title: An Open-label, Multicentre, Single-arm Trial of Monthly Injections of Depot Buprenorphine in People With Opioid Dependence
Brief Title: Community Studies of Long Acting Buprenorphine (CoLAB)
Acronym: CoLAB
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Marianne Byrne, Clinical Trials Manager, National Drug and Alcohol Research Centre, The University of New South Wales
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CoLAB1801
Record Dates: First submitted 2019-01-16; First posted 2019-01-18 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Sublocade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Depot buprenorphine arm (Experimental): All participants will receive monthly injections of depot buprenorphine (RBP-6000, Sublocade)
  Interventions: Drug: RBP-6000

INTERVENTIONS:
Drug: RBP-6000 — All study participants are scheduled to receive monthly subcutaneous injections of depot BPN, RBP-6000. RBP-6000 (BPN in the ATRIGEL® Delivery System) contains buprenorphine (200mg/mL) in the ATRIGEL® Delivery System, which provides sustained plasma level of BPN over a minimum of 28 days.
  Other Names: Sublocade

SUMMARY:
Despite research demonstrating the efficacy of buprenorphine (BPN), effectiveness in real-world settings has been limited by shorter retention than for methadone, and the need for daily or near-daily dosing (frequently supervised in Australia). Newly developed sustained-release BPN formulations could provide rapid onset and sustained release of BPN.

Current formulations include six-monthly implants, and once-weekly or once-monthly injections, removing the need for frequent clinic or pharmacy attendance. Improved medication adherence may result in improved patient outcomes and fewer unintended consequences such as diversion, but more data are needed in real-world settings. These innovations have the potential to dramatically change the treatment settings and options for people who are opioid dependent.

The study aims to evaluate the patient outcomes following the implementation of a monthly BPN depot injection for the treatment of opioid dependence in community-based treatment settings with a focus on opioid and other illicit drug use, adherence and retention, and participants' experiences of the implementation.

DETAILED DESCRIPTION:
Opioid agonist treatment (OAT) is effective for opioid dependence and newer extended-release buprenorphine (BUP-XR) injections represent a significant development. The Community Long-Acting Buprenorphine (CoLAB) study aims to evaluate client outcomes among people with opioid dependence receiving 48 weeks of BUP-XR treatment, and examines the implementation of BUP-XR in diverse community healthcare settings in Australia.

The CoLAB study is a prospective single-arm, multicentre, open-label trial of monthly BUP-XR injections in people with opioid dependence. Participants are being recruited from a network of general practitioner and specialist drug treatment services located in the states of New South Wales, Victoria and South Australia in Australia. Following a minimum 7 days on 8-32mg of sublingual buprenorphine (+/- naloxone), participants will receive monthly subcutaneous BUP-XR injections administered by a healthcare practitioner at intervals of 28 days (-2/+14 days). The primary endpoint is participant retention in treatment at 48 weeks after treatment initiation. Secondary endpoints will evaluate dosing schedule variations, craving, withdrawal, substance use, health and well-being, and client-reported treatment experience. Qualitative and costing sub-studies will examine implementation barriers and facilitators at the client and provider level.

ELIGIBILITY:
The study population is individuals diagnosed with opioid dependence who are currently receiving sublingual buprenorphine treatment at participating drug and alcohol services, express interest in receiving depot buprenorphine injections and are deemed suitable for treatment with RBP-6000 by the Investigator.

Inclusion criteria

To be eligible for the study, participants must meet all of the following inclusion criteria:

1. Voluntarily signed the informed consent form
2. Aged 18 to 65 years
3. Opioid-dependent (ICD-10) currently receiving treatment
4. Has been receiving 8-32mg sublingual buprenorphine +/- naloxone tablets/film for at least 7 days
5. Negative pregnancy test at screening and baseline in females of childbearing potential (please refer to Section 5.7 for long acting reversible contraceptive methods with efficacy considered to reasonably eliminate pregnancy potential)

Exclusion criteria

Participants who meet any of the exclusion criteria are not to be enrolled in this study:

1. Currently lactating or pregnant, or of childbearing potential and not willing to avoid becoming pregnant during the study
2. History or presence of allergic or adverse response (including rash or anaphylaxis) to buprenorphine or the ATRIGEL® Delivery System
3. Significant, medical or psychiatric conditions (other than opioid dependence), or other circumstances which, in the opinion of the Investigator, would compromise compliance with the protocol and/or patient safety. Specific conditions of interest include severe hepatic disease (Child-Pugh Class B), severe renal or respiratory disease, or severe cognitive impairment or psychiatric condition that impairs the ability to provide informed consent (e.g. psychosis, delirium, hypomania, severe depression or suicidal ideation)
4. Subjects who are currently participating in any other clinical study involving investigational medication(s)
5. Inability or unwillingness to provide informed consent or abide by the requirements of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-22 (Actual); Primary Completion 2020-11-01 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Participant retention | Retention in dosing schedule at 48 weeks
  To examine treatment retention at 48 weeks following initiation of monthly depot RBP-6000 buprenorphine injections in patients with opioid dependence transferred from a stable dose of sublingual buprenorphine.

SECONDARY OUTCOMES:
BUP-XR treatment retention and engagement in ongoing clinical care | 48 weeks
  To examine BUP-XR treatment retention and engagement in ongoing clinical care at 48 weeks ortion of participants retained in treatment at 48 weeks following initiation of monthly depot buprenorphine injections and engaged in ongoing clinical care. Treatment retention is defined as remaining on active depot buprenorphine medication AND completing a clinical assessment at 48 weeks.
Changes in opioid withdrawal | 48 weeks
  Change in opioid withdrawal assessed by clinical opioid withdrawal scale (COWS) and subjective opioid withdrawal scale (SOWS)
Changes in client-reported opioid craving | 48 weeks
  Change in client-reported opioid craving assessed by opioid craving scale
Changes in client-reported drug use | 48 weeks
  Change in client-reported use of opioids and other drugs, assessed by the Australian Treatment Outcomes Profile (ATOP) instrument
BUP-XR dosing schedule adherence | 48 weeks
  To evaluate client utilisation of buprenorphine medication during the study, including BUP-XR dose variation, adherence with dosing schedule, and dose supplementation
BUP-XR safety and tolerability | 48 weeks
  To evaluate treatment safety and tolerability by monitoring adverse events, and events of clinical interest such as drug-drug interactions and pain management in clients treated with BUP-XR
Changes in client-report pain and enjoyment | 48 weeks
  To describe client-reported changes to pain and enjoyment of life, assessed by the Pain, Enjoyment, General Activity (PEG) scale
Demographic factors associated with treatment retention | 48 weeks
  To evaluate demographic factors (gender, age, education) associated with treatment retention, assessed by demographic questionnaire
Client treatment satisfaction score | 48 weeks
  Client-reported treatment satisfaction assessed by the Treatment Questionnaire for Medication Satisfaction (TQSM)
BUP-XR treatment costs | 48 weeks
  Costs to services delivering BUP-XR assessed by site-reported expenses and time and motion study

CONTACTS AND LOCATIONS:
Overall Officials: Michael Farrell, Principal Investigator — National Drug and Alcohol Centre, University of New South Wales
Locations (6):
- Australia (6):
  - Drug and Alcohol Services, Hunter New England Local Health District, Newcastle, New South Wales
  - Drug and Alcohol Services, North Sydney Local Health District, Saint Leonards, New South Wales
  - Drug and Alcohol Services, South Australia (DASSA), Morphett Vale, South Australia
  - Western Health Drug Services, Footscray Hospital, Footscray, Victoria
  - Frankston Healthcare, Frankston, Victoria
  - Rankin Court Treatment Centre, St Vincent's Hospital Sydney, Darlinghurst

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Farrell M, Shahbazi J, Byrne M, Grebely J, Lintzeris N, Chambers M, Larance B, Ali R, Nielsen S, Dunlop A, Dore GJ, McDonough M, Montebello M, Nicholas T, Weiss R, Rodgers C, Cook J, Degenhardt L; CoLAB study team. Outcomes of a single-arm implementation trial of extended-release subcutaneous buprenorphine depot injections in people with opioid dependence. Int J Drug Policy. 2022 Feb;100:103492. doi: 10.1016/j.drugpo.2021.103492. Epub 2021 Nov 1. PMID 34736130
- [Derived] Larance B, Byrne M, Lintzeris N, Nielsen S, Grebely J, Degenhardt L, Shahbazi J, Shanahan M, Lancaster K, Dore G, Ali R, Farrell M; CoLAB study team. Open-label, multicentre, single-arm trial of monthly injections of depot buprenorphine in people with opioid dependence: protocol for the CoLAB study. BMJ Open. 2020 Jul 31;10(7):e034389. doi: 10.1136/bmjopen-2019-034389. PMID 32737087